CLINICAL TRIAL: NCT02248337
Title: Colon Cleasing for Colonoscopy in Patients With IBD Colitis: Efficacy and Acceptability of 4 Liter PEG vs 2 Liter PEG Plus Bisacodil
Brief Title: Low Volume Colon Preparation for IBD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Luigi Sacco University Hospital (Other)
Responsible Party: Principal Investigator, Gianpiero Manes, MD, Luigi Sacco University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LOVOL-IBD
Record Dates: First submitted 2014-09-20; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Inflammatory Bowel Disease
Keywords: Colon preparation; Colonoscopy; Inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 Liter PEG (Active Comparator): Colon preparation for colonoscopy: PEG 4 Liter before endoscopy
  Interventions: Drug: Colon preparation for colonoscopy
- 2 Liter PEG plus bisacodil (Experimental): Colon preparation for colonoscopy: PEG 2 L before endoscopy
  Interventions: Drug: Colon preparation for colonoscopy

INTERVENTIONS:
Drug: Colon preparation for colonoscopy — Colon cleansing prior to perform colonoscopy
  Other Names: Colon cleansing

SUMMARY:
Comparison of two PEG-based bowel cleansing regimens in patients with inflammatory bowel disease.

DETAILED DESCRIPTION:
Low-volume preparations are gaining attention for higher acceptability. This study compares efficacy, safety and tolerability of a 2L PEG solution plus bisacodil with a 4L PEG solution in patients with inflammatory bowel disease-related colitis.

This will be a multicenter, randomized, single-blind study. Adult outpatients with IBD colitis undergoing colonoscopy will receive either 2L PEG plus biscodil or 4L PEG. Bowel cleansing will be assessed using the Ottawa Scale and rated as adequate if <6. Patient acceptance, satisfaction, and related symptoms will be also recorded. The study will also focus on the factors affecting quality of preparation in inflammatory bowel disease patients such as disease characteristics and administration regimen

ELIGIBILITY:
Inclusion Criteria:

-Adult outpatiets with IBD colitis undergoing colonoscopy

Exclusion Criteria:

* Previous colon resection, ileus, intestinal obstruction, toxic megacolon, severe heart failure (NYHA Class III or IV), acute cardiovascular disease, uncontrolled arterial hypertension (systolic pressure >170 mmHg, diastolic pressure >100 mmHg), severe liver cirrhosis (Child-Pugh score C) or renal failure (creatinine clearance<30 mL/minute), ascites, phenylketonuria, and glucose-6-phosphate dehydrogenase deficiency
* Pregnant or breastfeeding women were also excluded

Ages: 18 Years to 85 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Efficacy | During endoscopy within 24 hours after preparation
  Quality of colon cleansing assesse with Ottawa bowel preparation score

SECONDARY OUTCOMES:
Compliance | during product assumption
  Intake of at least 75% of the product volume
Tollerability | during product assumption
  Occurrence of discomfort during drug intake
safety | From drug intake to the end of colonoscopy
  Occurrence of side effects

CONTACTS AND LOCATIONS:
Overall Officials: gianpiero manes, MD, Study Chair — AO G. Salvini Garbagnate Milanes
Locations (1):
- Luigi Sacco University Hospital, Milan, Italy

REFERENCES:
- [Derived] Manes G, Fontana P, de Nucci G, Radaelli F, Hassan C, Ardizzone S. Colon Cleansing for Colonoscopy in Patients with Ulcerative Colitis: Efficacy and Acceptability of a 2-L PEG Plus Bisacodyl Versus 4-L PEG. Inflamm Bowel Dis. 2015 Sep;21(9):2137-44. doi: 10.1097/MIB.0000000000000463. PMID 26164666